CLINICAL TRIAL: NCT05271422
Title: A Single Center, Single-blind, Exploratory Study to Evaluate the Efficacy and Safety of the Application of Pulse Electrical Stimulation Around Eye in Dry Eye Disease Patients Who Are Scheduled for LASEK Surgery
Brief Title: Application of Pulse Electrical Stimulation Around Eye in Dry Eye Disease Patients Scheduled for LASEK Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nu Eyne Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NE_DED_001
Record Dates: First submitted 2022-02-25; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Dry eye disease patients (n=12)
  Interventions: Device: Real Pulse Electrical Stimulation (NuEyne 01)
- Control Group (Sham Comparator): Dry eye disease patients (n=12)
  Interventions: Device: Sham Pulse Electrical Stimulation

INTERVENTIONS:
Device: Real Pulse Electrical Stimulation (NuEyne 01) — Patients wear our clinical trial device 15~30 mins once a day for 14 days and once a week from the 15th day to the 12th week.
  Arms: Experimental Group
Device: Sham Pulse Electrical Stimulation — Patients wear our clinical trial device 15~30 mins once a day for 14 days and once a week from the 15th day to the 12th week.
  Arms: Control Group

SUMMARY:
This study aims to evaluate the efficacy and safety of applying pulse electrical stimulation around eye in dry eye disease patients who are scheduled for LASEK surgery.

DETAILED DESCRIPTION:
Duration of study period (per participant): Screening period (0-14 days), Intervention period (12 weeks), F/U period (2 weeks) Patient needs to visit site at least 9 times (Screening, baseline, V1, V2, V3, Tele-visit, V4, V5, F/U Tele-visit). Baseline visit will be done on the day of surgery. Visit 1, 2, 3, Tele-visit, 4, 5, F/U Tele-visit is 1 day, 3 days, 1 weeks, 2 weeks, 4 weeks, 12 weeks and 16weeks after baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 19 to 60 years of age, at the time of screening
* Those who are scheduled to get LASEK surgery
* According to the guidelines for diagnosing dry eye syndrome of Korean Corneal Disease Study Group, those who fall under Grade II or higher
* Those with an OSDI score of 13 or higher
* A person who has no pregnancy plan during the clinical trial period and has agreed to an effective contraceptive plan for Women of child bearing potential (WOCBP) by a doctor
* A person who voluntarily agreed to participate in this clinical trial

Exclusion Criteria:

Patients who meet any of the exclusion criteria are excluded from this clinical trial.

* A person with an uncontrollable systemic chronic disease (diabetes mellitus)
* Those who are allergic to drugs such as Fluorescein Solution or ophthalmic anesthetics
* In a case where there is a history of receiving ophthalmic surgery known to affect the tear layer within the last 6 months (e.g., Cataract, Pterygium surgery)
* A person who takes systemic drugs (e.g., tetracycline derivatives, antihistamine, isotretinoin)
* A person who has eyelid diseases or structural abnormalities
* A person with acute eye infection or inflammation of the eyeball not related to Meibomian gland dysfunction
* A person with abnormalities in the eyelids or eyelashes
* A person with an eye condition or ophthalmic disease that is considered unsuitable for surgery (e.g., detachment of the retina, cataract)
* Pregnant or lactating women
* Those who can't understand or read the consent form of this clinical trial (e.g., illiterate or foreigners)
* Any other cases that PI considers hard to participate in this clinical trial (e.g., heart-related problems, seizure, epilepsy. Patients transplanted metal or electronic device in head & neck. Patient suffering from unknown pain. Patients who are warned not to use our clinical trial device or is prohibited from using it (e.g., pacemaker user).)

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Changes in Ocular Surface Disease Index (OSDI) score | baseline, 1, 4, 12 weeks
  Check the changes in Ocular Surface Disease Index (OSDI) score
Changes in Tear break-up time (T-BUT) | Time Frame: baseline, 1, 4, 12 weeks
  Check the changes in Tear break-up time (T-BUT)

SECONDARY OUTCOMES:
Changes in 5-Item Dry Eye Questionnaire (DEQ-5 score) | baseline, 1, 4, 12 weeks
  Check the changes in 5-Item Dry Eye Questionnaire (DEQ-5 score)
Changes in Patient Evaluation of Eye Dryness (SPEED) II questionnaire score | baseline, 1, 4, 12 weeks
  Check the changes in Patient Evaluation of Eye Dryness (SPEED) II questionnaire score
Changes in Visual Analogue Scale (VAS) score | baseline, 1 day, 3 days, 7 days
  Check the changes in Visual Analogue Scale (VAS) score
Changes in Staining Score | baseline, 1, 4, 12 weeks
  Check the changes in Staining Score
Changes in Matrix Metalloproteinase-9 (MMP-9) level | baseline, 4, 12 weeks
  Check the changes in Matrix Metalloproteinase-9 (MMP-9) level
Changes in LipiView Eye Lipid Layer Thickness | baseline, 4, 12 weeks
  Check the changes in LipiView Eye Lipid Layer Thickness
Changes in Tear Volume | baseline, 1, 4, 12 weeks
  Check the changes in Tear Volume
Changes in Tear Osmolarity | baseline, 4, 12 weeks
  Check the changes in Tear Osmolarity
Changes in the length of the aesthesiometer's filament in centimeters | baseline, 1, 4, 12 weeks
  Check the changes in the length of the aesthesiometer's filament in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Donghui Lim, Ph. D., MD., Principal Investigator — Department of Ophthalmology, Samsung Medical Center
Locations (1):
- Department of Ophthalmology, Samsung Medical Center, Seoul, South Korea